CLINICAL TRIAL: NCT07056933
Title: Effect of Minoxidil Solution Iontophoresis on Androgenic Alopecia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim Mohammed Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/005693
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minoxidil-treated scalp (Experimental): 5% minoxidil through iontophoresis will be applied to one half of the scalp twice daily at home.
  Interventions: Other: Minoxidil solution iontophoresis
- Saline-treated scalp (Active Comparator): The other half of the scalp will receive a placebo solution, (eg saline) with current application.
  Interventions: Other: saline solution iontophoresis

INTERVENTIONS:
Other: Minoxidil solution iontophoresis — The half of the scalp of the participants will be treated with 5% minoxidil solution through Iontophoresis that will be applied at small low voltage (typically 10 V or less) continuous constant current (typically 0.5 mA/cm2 or less) to push a charged drug into skin or other tissue, twice daily at home.
  Arms: Minoxidil-treated scalp
Other: saline solution iontophoresis — The other half of the scalp of the participants will be treated with placebo saline solution ( control) with the current application.
  Arms: Saline-treated scalp

SUMMARY:
The aim of the study is to evaluate the therapeutic efficiency of minoxidil solution iontophoresis on Androgenic Alopecia.

DETAILED DESCRIPTION:
Hair is an important component of identity and self-image. Hair loss can lead to a variety of psychological difficulties and have a negative impact on quality of life (QoL). Loss of self-confidence lowered self-esteem, and heightened self-consciousness are common responses to hair loss, particularly for women. People with alopecia are more likely to develop depression and anxiety.

Some studies have proposed iontophoresis and ultrasound as energetic drug delivery methods to favor topical therapy of alopecia. Iontophoresis is a non-invasive technique that applies a small electric current (of no more than 0.5 mA/cm2) on the skin's surface to increase and control drug delivery. The technique is widely studied to stimulate the skin penetration and permeation of hydrophilic drugs, which would not be absorbed by the skin when passively applied. The transport of drugs through the skin as a result of the electric current is driven by two different mechanisms, ie, electromigration in the case of charged drugs and electroosmosis in the case of neutral drugs.

Furthermore the need of this study is developed from the lack in quantitative knowledge and information in published studies which investigate effect of minoxidil solution iontophoresis on Androgenic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-five adult aged 18-65 with diagnosed androgenic alopecia.
* They diagnosed as Androgenic alopeacia by their physicians and referred for physical therapy management.
* Medically and psychologically stable patients.

Exclusion Criteria:

* History of hypersensitivity to minoxidil solution or Intophoresis.
* Scalp infection
* Concurrent hair loss treatments.
* Patients who suffer from hypertrophic and/or keloidal scars and a skin condition in the area of Androgenic alopecia that would interfere with study procedures.
* plaque psoriasis, tattoo, birthmark, facial hair.
* Patients with medical red flags as severe psychiatric disorder or cognitive deficits.
* Medically unstable and uncooperative patients.
* Immunocompromised status.
* History of skin cancer.
* Recurrent herpes viral infection.
* Pregnancy or breastfeeding status.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2025-07-08 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the number of hair follicles | 12 weeks
  Trichoscopy will be used to detect the change in the number of hair follicles as a comparison between before and after intervention. Trichoscopy helped with the definitive diagnosis of Alopeacia in patients for whom the clinical diagnosis was doubtful, which was confirmed by histopathology. Thus trichoscopy is a noninvasive, sensitive and specific investigation that is valuable in women with alopecia, the cause of which is otherwise very difficult to assess clinically, and it has a definite role in the diagnosis of cases with an atypical clinical picture.Trichoscopy results were obtained in frontal, occipital and both temporal areas of scalp, including number of yellow dots and vellus hairs, number of hairs in one pilosebaceous unit and percentage of follicular ostia with perifollicular hyperpigmentation.

SECONDARY OUTCOMES:
Change of hair thickness | 12 weeks
  Global Photographic System will be used to detect the change of hair thickness as a comparison between before and after intervention.
  The Global Photographic Assessment is useful for determining overall clinical changes in a patient over times period in a standardized manner, Global Photographs are head shots taken a short distance away from the patients, a patient is usually photographed from the front, top, sides, and back to show accordingly a frontal hair line, crown, partition and vertex.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Abdelgayed, Study Director — Cairo University; Amal Abd Elbaky, Professor, Study Chair — Cairo University
Locations (1):
- Mahmoud Ibrahim Mohamed, Zagazig, Egypt